CLINICAL TRIAL: NCT02709343
Title: Phase 2 Randomised Controlled Trial of Bone-marrow Derived Mesenchymal Stromal Cells (MSC) for New Onset Chronic Lung Allograft Dysfunction (CLAD)
Brief Title: Trial of Bone-marrow Derived Mesenchymal Stromal Cells (MSC) for New Onset Chronic Lung Allograft Dysfunction
Acronym: ASSIST-CLAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Isopogen (Unknown); Cell and Tissue Therapies (Unknown)
Responsible Party: Principal Investigator, Daniel Chambers, A/Prof Daniel Chambers, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASSIST-CLAD
Record Dates: First submitted 2016-03-01; First posted 2016-03-16 (Estimated); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Chronic Lung Allograft Dysfunction (CLAD)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone-marrow derived MSCs (Experimental): 4 doses of Allogeneic bone-marrow derived MSCs (2x106 cells/kg) given intravenously twice weekly for 2 weeks
  Interventions: Drug: Bone-marrow derived MSCs
- Placebo (Placebo Comparator): Placebo product manufactured to look like MSCs
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bone-marrow derived MSCs — Allogeneic ex vivo expanded, bone marrow-derived mesenchymal stromal cells
  Other Names: MSC
  Arms: Bone-marrow derived MSCs
Drug: Placebo — Placebo product visually very similar to mesenchymal stromal cells
  Arms: Placebo

SUMMARY:
This study is designed for lung transplant patients who have developed chronic lung allograft dysfunction (CLAD). Consented patients will receive 4 intravenous doses of allogeneic, bone-marrow-derived MSCs (2*10^6 cells/kg/dose) or matching placebo over a period of 2 weeks with a 12 month follow up.

DETAILED DESCRIPTION:
This is a phase 2, multi-center, randomized study (n=82, 1:1 MSC:placebo) where consented patients will receive 4 intravenous doses of IMP over a period of 2 weeks. Patients must provide written informed consent and meet the all Inclusion Criteria and none of the Exclusion Criteria to be eligible. Screening procedures include obtaining medical history, current medications, questionnaires, vital signs, Chest Xray, 6 Minute walk test and blood tests. Historical chest CT and full lung function from 12 weeks prior to screening may be used. Bronchoscopy with biopsy must have been performed no more than 6 months prior to screening. A bronchoscopy with bronchoalveolar lavage (BAL) is required, however will not need to be repeated if performed within 14 days prior to the baseline visit. Patients will then receive 4 infusions of MSC/placebo over a period of 2 weeks, with follow up at Week 3,6,10,14,28,41 and week 54.

ELIGIBILITY:
Inclusion Criteria:

1. Bilateral lung transplant recipients aged ≥ 18 years and at least 6 months post-transplant. Patients with other organs transplanted (eg heart, liver, kidney) or those who have undergone lobar transplantation, or re-transplantation, are potentially eligible.
2. New-onset CLAD (defined as a persistent (3weeks apart) fall in FEV1 of at least 20% from the mean of the two best post-transplant values taken at least 3 weeks apart) in the 12 months prior to the screening visit. Other causes of a fall in FEV1 (acute cellular or humoral rejection, active infection, anastomotic stenosis etc.) must be excluded as per international guidelines.
3. Stable immunosuppression regimen, as assessed by the investigator, in the 8 weeks prior to the screening visit.
4. Available for all specified assessments at the study site through the completion of the study, including the protocol bronchoscopies.
5. Provision of written informed consent.

Exclusion Criteria:

1. Any condition that in the opinion of the Investigator may interfere with the safety of the patient, his / her completion of required follow-up visits or evaluation of the study objectives
2. Untreated cellular or humoral rejection
3. Clinically meaningful and untreated viral, bacterial or fungal infection
4. Use of azithromycin or another macrolide antibiotic, if commenced within 8 weeks of the screening visit
5. Intravenous pulsed methylprednisolone, within 4 weeks of the screening visit
6. Use of extracorporeal photopheresis, within 4 weeks of the screening visit
7. Use of total lymphoid irradiation, within 4 weeks of the screening visit
8. Poor functional status not expected to survive 6 months
9. Allergy to beef products
10. Women who are pregnant, breast-feeding or unwilling to use adequate contraception
11. Patients who are currently participating in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From baseline to week 54
  Progression-free survival is a composite end-point of freedom from CLAD progression or death from any-cause. CLAD progression is defined as fall in FEV1 > 10% from the baseline (screening visit) FEV1 to the 12 month (week 54) visit.

SECONDARY OUTCOMES:
Time to fall in FEV1 > 10% | From the baseline (screening) visit
  Defined as fall in FEV1 > 10% from the baseline (screening visit) FEV1
Freedom from Bronchiolitis Obliterans Syndrome (BOS) grade 3 | Week 54
  BOS grade 3 is defined as FEV1 <50% of the best-post-transplant FEV1
All cause mortality | Week 54
CLAD-specific mortality | Week 54
  Defined as any death felt by the investigator to be at least partially related to CLAD.
Freedom from acute rejection | From baseline to week 54
  Acute rejection defined as any biopsy proven episode of acute vascular (A1-A4) or airway (B1R or B2R) rejection.
Freedom from the development of new donor specific anti-HLA antibodies | From baseline to week 14
  An anti-HLA antibody (any mean fluorescent intensity level) with specificity for a donor HLA type at 3 months which was not present prior to IMP treatment
Freedom from CLAD progression | From baseline to week 54
  CLAD progression is defined as fall in FEV1 > 10% from the baseline (screening visit) FEV1 at 12 months.
Rate of FEV1 decline | From baseline to week 54
  Rate of FEV1 decline is defined as the slope of the regression line for FEV1 between the screening visit and week 54
Rate of FVC decline | From baseline to week 54
  Rate of FVC decline is defined as the slope of the regression line for FVC between the screening visit and week 54
Change in 6-minute walk distance (6MWD) | From baseline to week 54
  Change in 6MWD is defined as the difference between the 6MWD at screening and the week 54 visit. Patients who have died by week 54 will receive a 6MWD of 0.
Change in St George's Respiratory Questionnaire (SGRQ) Score | From baseline to week 54
  Change in SGRQ is defined as the difference between the total SGRQ at screening and the week 54 visit. Patients who have died by week 54 will receive a SGRQ of 0.
Inpatient bed-days | From baseline to week 54
  This is defined as the aggregate of inpatient bed-days between the screening visit and week 54.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Chambers, MBBS MD, Principal Investigator — University of Queensland & The Prince Charles Hospital
Locations (5):
- Australia (5):
  - St Vincents Hospital, Sydney, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be analysed and shared with collaborators with the plan to publish the results.